CLINICAL TRIAL: NCT02204566
Title: Pilot Study of OFDI Capsule Imaging of the Esophagus of Patients With Atrial Fibrillation Following RF Ablation
Brief Title: OFDI Capsule Imaging in Patients With Atrial Fibrillation Undergone Radio Frequency (RF) Ablation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Guillermo Tearney, Professor of Pathology, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 2012-P-001952; 5R01CA103769-08 (NIH)
Record Dates: First submitted 2014-06-17; First posted 2014-07-30 (Estimated); Results first posted 2019-08-26 (Actual); Last update posted 2019-11-08 (Actual); Status verified 2019-10

CONDITIONS: Atrial Fibrillation
Keywords: OFDI; RF Ablation; Atrial Fibrillation; Imaging; Esophagus
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OFDI Capsule Imaging (Experimental): Subject will swallow the OFDI capsule and imaging will be acquired using the OFDI Imaging system.
  Interventions: Device: OFDI Capsule

INTERVENTIONS:
Device: OFDI Capsule — Imaging of the esophagus using the OFDI Capsule and system

SUMMARY:
12 patients with Atrial Fibrillation, a kind of irregular heart beat who have undergone Radio frequency (RF) ablation will be asked to swallow the capsule.

As they swallow the capsule, images of the esophagus will be taken to see if the RF ablation caused any form of damage to the esophagus considering it being so close to the heart.

After the capsule has been removed from the mouth, they will be asked about the tolerability of the capsule.

DETAILED DESCRIPTION:
A total of 12 patients with a known diagnosis of Atrial Fibrillation who have previously undergone Atrial RF ablation will be enrolled in the study. Patients will be asked to swallow the OFDI capsule while being unsedated. The capsule is attached to a tether that allows the capsule operator to navigate the capsule as it progresses down the esophagus using natural propulsion called peristalsis as well as to bring it back up to pulled out of the mouth when the procedure is done.

As the capsule progresses down the esophagus, multiple, two dimensional, microscopic cross- sectional images of the esophagus are acquired.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be over 18 years of age
* Subjects must be able to give informed consent.
* Subjects must be referred to Massachusetts General Hospital (MGH) endoscopy for RF Ablation treatment of their Atrial Fibrillation.

Exclusion Criteria:

* Subjects with current esophageal strictures and dysphagia
* OR subjects with a prior history of intestinal strictures, prior GI surgery or intestinal Crohn's disease.
* OR subjects with a known history of chronic aspiration.
* OR women who are currently pregnant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Guillermo Tearney, MD., PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | OFDI Capsule Imaging
Started | 5
Completed | 1
Not Completed | 4

BASELINE CHARACTERISTICS:
Arm/Group | OFDI Capsule Imaging
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62 (7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Feasibility of a Tethered OFDI Capsule in Patients With Atrial Fibrillation Following RF Ablation That Swallow the OFDI Capsule
Description: An investigator will assess the quality of the recorded images and movies obtained with each exam after the imaging is completed. A total of 6 subjects were enrolled in this study. 1 participant was not analyzed as they could not attempt to swallow the capsule.
Time Frame: After the completed imaging session
Measure: Count of Participants; unit: Participants
Groups:
- Feasibility: Number of Participants with Acceptable Quality of Images Who Swallow the OFDI Capsule
Arm/Group | Feasibility
Number analyzed (Participants) | 5
Participants | 1

ADVERSE EVENTS:
Arm/Group | OFDI Capsule Imaging
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No